CLINICAL TRIAL: NCT03378362
Title: A Prospective Study on Pain Relief and Functional Outcome After Partial Denervation of the Wrist
Brief Title: Pain Relief and Functional Outcome After Partial Denervation of the Wrist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Elin Swärd, MD, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Karolinska Institute
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Wrist Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Partial denervation of the wrist joint (Experimental): Patients will be operated with a partial denervation of the wrist through a single dorsal approach.
  Interventions: Procedure: Partial denervation of the wrist joint

INTERVENTIONS:
Procedure: Partial denervation of the wrist joint — Partial denervation of the wrist (posterior and anterior interosseous neurectomy) through a single dorsal approach.

SUMMARY:
Prospective study on the effect of partial wrist denervation (ie combined anterior and posterior interosseous neurectomy) on pain relief on functional outcome in patient with wrist osteoarthritis. The impact of psychological factors on postoperative outcome will be studied.

ELIGIBILITY:
Inclusion criteria

1. Chronic wrist pain (≥6 months) due to posttraumatic arthritis after distal radius fracture or SLAC/SNAC arthritis or arthritis due to Mb Preiser/Mb Kienböck where surgical unloading of the bone isn't possible.
2. Pain is refractory to nonsurgical management such as bracing, corticosteroid injection, oral analgesics, NSAIDs, physiotherapy.

Exclusion criteria

1. Rheumatoid or other inflammatory arthritis.
2. Previous wrist surgery with simultaneous PIN/AIN neurectomy.
3. Simultaneous arthritis or symptomatic instability of the distal radio ulnar (DRU) joint on the ipsilateral side.
4. Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction).
5. Patient's wish for a definite procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-31 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Disability of the Arm, Shoulder and Hand score (DASH) | peroperatively, 3, 6 and 12 months postoperatively
  questionnaire

SECONDARY OUTCOMES:
Change in Patient Related Wrist Evaluation (PRWE) | peroperatively, 3, 6 and 12 months postoperatively
  questionnaire
Change in EQ5D | peroperatively, 3, 6 and 12 months postoperatively
  questionnaire
Change in Hospital Anxiety and Depression Scale (HADS) | peroperatively, 3, 6 and 12 months postoperatively
  questionnaire. Determines the levels of anxiety and depression. 14 item scale that generates ordinal data. Seven items relate to anxiety and seven to depression. Each item is scored from 0-3, which means that a person can score between 0-21 for either depression or anxiety. A score of 11 or above on either scale in considered to repressent depression or anxiety.
Change in range of motion, grip strength | peroperatively, 3, 6 and 12 months postoperatively
  objective physical function
Change in Sence Of Coherence -13 (SOC13) | peroperatively, 3, 6 and 12 months postoperatively
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wilcke, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Handkirurgiska kliniken Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided